CLINICAL TRIAL: NCT05353894
Title: Effect of Food and Formulation on the Pharmacokinetics, Safety, and Tolerability of GNS561 After One Single Dose (50 and 200mg) in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Genoscience Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GNS561-CL-I-Q-0321
Record Dates: First submitted 2022-04-14; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 Cohort 1 (Experimental): Three (3) Healthy volunteers, each receiving a single oral dose (50mg) of GNS561 tablets and capsules, after a high fat meal and with a wash-out period of seven days.
  Interventions: Drug: GNS561 oral tablets and capsules
- Part 1 Cohort 2 (Experimental): Six (6) healthy volunteers, each receiving a single oral dose (200mg) of GNS561 tablets and capsules, after a high fat meal and with a wash-out period of fourteen days.
  Interventions: Drug: GNS561 oral tablets and capsules
- Part 2 (Experimental): Nine (9) healthy volunteers, each receiving a single oral dose (200mg) of GNS561 tablets or capsules (according results of Part 1), in fed condition then in fasting condition, after a wash-out period of fourteen days.
  Nine (9) other healthy volunteers, each receiving a single oral dose (200mg) of GNS561 tablets or capsules (according results of Part 1), in fasting condition then in fed condition, after a wash-out period of fourteen days.
  Interventions: Drug: GNS561 oral tablets and capsules

INTERVENTIONS:
Drug: GNS561 oral tablets and capsules — Two formulations and Two dosage will be compared

SUMMARY:
GNS561 is a drug used in preliminary phase 1b study for treatment of patients with primary and secondary liver cancer. The formulation used was oral capsule.The objective of this study in healthy volunteers is to compare pharmacokinetics, safety and tolerability of different formulations (tablets and capsules) and dosage (50 and 200mg) of GNS561 after single oral administration in first part and to evaluate the food effect on pharmacokinetics in second part.

ELIGIBILITY:
Inclusion Criteria:

* BMI will be between 18 (inclusive) and 26 kg/m² (inclusive).
* Participants must be in good general health, with no significant medical history, have no clinically significant (CS) abnormalities on physical examination, vital signs, and 12-lead ECG at Screening and/or before administration of the first dose of study drug
* Have a Fridericia's correction factor for QT (QTcF) ≤ 450 ms for male participants and ≤ 470 ms for female participants on 12-lead ECG
* Women subjects of childbearing potential must have a negative serum/urine pregnancy test at screening and baseline
* Women subjects of childbearing potential and male subjects must agree to use adequate highly effective contraception for the duration of study participation and up to 6 months following completion of therapy
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Able to understand and provide written informed consent.

Exclusion Criteria:

* Pregnant or breast-feeding mothers
* Known allergic reaction to quinolone derivatives (e.g., quinine, choloroquine, mefloquine)
* Subjects with any clinically significant laboratory abnormality
* History of QT prolongation (QTc ≥ 500 ms) or family history of long QT arrythmia or cardiac disease or bradycardia < 50/mn or uncorrected hypokalemia
* On going uncontrolled infection disease
* History of pre-existing retinopathy or maculopathy
* Participation in any investigational clinical investigation ≤ 4 weeks prior to first planned dose of GNS561
* Malabsorption issues (e.g., gastric bypass or gastrectomy patients), current or history significant gastrointestinal diseases
* Patient with a mental or legal disability

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-05-02 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | from first administration until 29 days
  adverse events
Maximum Plasma Concentration (Cmax) | Day 1, Day 2, Day 3, Day 4 and Day 7
  blood samples at different time from GNS561 administration

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Day 1, Day 2, Day 3, Day 4 and Day 7
  blood samples at different time from GNS561 administration

CONTACTS AND LOCATIONS:
Locations (1):
- Genoscience Pharma, Marseille, France

IPD SHARING:
Plan to Share IPD: No